CLINICAL TRIAL: NCT03704818
Title: Evaluating the Effect of Dapagliflozin, an SGLT-2 Inhibitor, on the Counterregulatory Response to Hypoglycemia in Individuals With Type 1 Diabetes
Brief Title: Dapagliflozin Effects on Hypoglycemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UC-MEDJP-01
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin 5mg (Experimental)
  Interventions: Drug: Dapagliflozin 5mg
- Placebo (Experimental)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin 5mg — Dapagliflozin treatment taken daily for 4-weeks.
  Other Names: Farxiga
  Arms: Dapagliflozin 5mg
Drug: Placebo Oral Tablet — Placebo treatment taken daily for 4-weeks.
  Arms: Placebo

SUMMARY:
The purpose of this research study will be to test and evaluate if dapagliflozin has an effect on the amount of glucagon (a hormone produced by the pancreas and stomach that stimulates liver glucose production) produced by the body and if that change will improve recovery time from hypoglycemia (low blood sugar) in participants with Type 1 Diabetes.

DETAILED DESCRIPTION:
The purpose of this research study will be to test and evaluate if dapagliflozin has an effect on the amount of glucagon (a hormone produced by the pancreas and stomach that stimulates liver glucose production) produced by the body and if that change will improve recovery time from hypoglycemia (low blood sugar) in participants with Type 1 Diabetes. The study is a blinded, placebo-controlled, crossover design, where participants will receive dapagliflozin during one treatment period and placebo during a separate treatment period with neither the study team nor participants knowing what they are receiving at any given time. Participants will have 9 clinic visits over the course of 14-16 weeks, with 3 of those visits being overnight stays. The overnight stays are intended to control blood sugars in a normal state throughout the night and then participants will complete a hypoglycemic challenge the following morning. The body's response to the hypoglycemic challenge will provide the information needed to determine if dapagliflozin had an effect on recovery time from hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent by the date of Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation
2. Male or female patient receiving insulin for the treatment of documented diagnosis of T1DM for at least 1 year at the time of Visit 1
3. Non-fasting C-peptide < 0.7 ng/mL at Visit 1
4. HbA1c ≤ 10.0% at Visit 1
5. Based on the Investigator's judgment patient must have a good understanding of his/her disease and how to manage it, and be willing and capable of performing the following study assessments (assessed at Visits 1):

   * patient-led management and adjustment of insulin therapy
   * reliable approach to insulin dose adjustment for meals, such as carbohydrate counting
   * reliable and regular home-based blood glucose monitoring
   * be able to perform ketone sample measurement when feeling ill and/or nauseated
   * implementation of an established "sick day" management regimen
6. Age ≥ 18 and ≤ 70 years at Visit 1
7. Body Mass Index (BMI) of 18.5 kg/m2 to 35.0 kg/m2 at Visit 1
8. eGFR ≥ 60 mL/min/1.73m²
9. Patients must be able and willing to perform study assessments

Exclusion Criteria:

1. History of T2DM, maturity onset diabetes of the young (MODY), pancreatic surgery or chronic pancreatitis
2. Pancreas, pancreatic islet cells or renal transplant recipient
3. T1DM treatment with any other antihyperglycemic drug (e.g. metformin, alpha- glucosidase inhibitors, SGLT-2 inhibitors, pramlintide, inhaled insulin, pre-mixed insulins, etc.) within 30 days of run-in (visit 2)
4. Occurrence of severe hypoglycemia involving coma and/or seizure that required hospitalization or hypoglycemia-related treatment by an emergency physician or paramedic within 3 months prior to Visit 1 or Visit 2
5. Occurrence of DKA within 3 months prior to Visit 1 or Visit 2
6. Acute coronary syndrome (non-STEMI, STEMI and unstable angina pectoris), stroke or transient ischemic attack (TIA) within 3 months prior to Visit 1 or Visit 2
7. Indication of liver disease, defined by serum levels of either alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase above 3 x upper limit of normal (ULN) at Visit 1
8. Current signs and symptoms of anemia accompanied by a hemoglobin laboratory value at or below 10.0 g/dL at screening.
9. Eating disorders such as bulimia or anorexia nervosa
10. Treatment with systemic corticosteroids within 30 days of run-in (visit 2), or planned initiation of such therapy at Visit 1 or Visit 2. Inhaled or topical use of corticosteroids (e.g. for asthma/chronic obstructive pulmonary disease) is acceptable.
11. Medical history of cancer or treatment for cancer in the last five years prior to Visit 1. Resected basal cell carcinoma considered cured is exempted.
12. Women who are pregnant, nursing, or who plan to become pregnant while in the trial
13. Intake of an investigational drug in another trial within 30 days prior to Visit 1
14. Patient not able to understand and comply with study requirements, based on Investigator's judgment
15. Any other clinical condition that, based on Investigator's judgment, would jeopardize patient safety during trial participation or would affect the study outcome (e.g. immunocompromised patients who might be at higher risk of developing genital or mycotic infections, patients with chronic viral infections etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Glucagon Response to Hypoglycemia | 12 Weeks
  Participants will undergo a baseline hypoglycemic clamp during which glucagon will be measured. Follow-up hypoglycemic clamps will be performed after each 4-week treatment period re-assessing glucagon.
Epinephrine Response to Hypoglycemia | 12 Weeks
  Participants will undergo a baseline hypoglycemic clamp during which epinephrine will be measured. Follow-up hypoglycemic clamps will be performed after each 4-week treatment period re-assessing epinephrine.
Norepinephrine Response to Hypoglycemia | 12 Weeks
  Participants will undergo a baseline hypoglycemic clamp during which norepinephrine will be measured. Follow-up hypoglycemic clamps will be performed after each 4-week treatment period re-assessing norepinephrine.
Cortisol Response to Hypoglycemia | 12 Weeks
  Participants will undergo a baseline hypoglycemic clamp during which cortisol will be measured. Follow-up hypoglycemic clamps will be performed after each 4-week treatment period re-assessing cortisol.
Growth Hormone Response to Hypoglycemia | 12 Weeks
  Participants will undergo a baseline hypoglycemic clamp during which growth hormone will be measured. Follow-up hypoglycemic clamps will be performed after each 4-week treatment period re-assessing growth hormone.
Hypoglycemia Awareness | 12 Weeks
  Participants will undergo a baseline hypoglycemic clamp during which they will complete the Edinburgh Hypoglycemia Scale (EHS). Follow-up hypoglycemic clamps will be performed after each 4-week treatment period re-assessing the EHS.
Trails Making B Performance Response to Hypoglycemia | 12 Weeks
  Participants will undergo a baseline hypoglycemic clamp during which they will complete the cognitive test, Trails Making B. Follow-up hypoglycemic clamps will be performed after each 4-week treatment period re-assessing Trails Making B.
Digit Symbol Substitution Performance Response to Hypoglycemia | 12 Weeks
  Participants will undergo a baseline hypoglycemic clamp during which they will complete the cognitive test, Digit Symbol Substitution. Follow-up hypoglycemic clamps will be performed after each 4-week treatment period re-assessing Digit Symbol Substitution.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boeder SC, Gregory JM, Giovannetti ER, Pettus JH. SGLT2 Inhibition Increases Fasting Glucagon but Does Not Restore the Counterregulatory Hormone Response to Hypoglycemia in Participants With Type 1 Diabetes. Diabetes. 2022 Mar 1;71(3):511-519. doi: 10.2337/db21-0769. PMID 34857545